CLINICAL TRIAL: NCT03834766
Title: Amphetamine Extended-Release Tablets in the Treatment of Adults With ADHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tris Pharma, Inc. (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRI108-ADD-400
Record Dates: First submitted 2019-02-04; First posted 2019-02-08 (Actual); Results first posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2019-12

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind (DB), placebo-controlled, parallel study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: AMPH ER Tab 5, 10, 15 & 20 mg Vs. Matching Placebo
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AMPH ER Tab (Active Comparator): Amphetamine Extended Release Tablets 5, 10, 15 and 20 mg
  Interventions: Drug: AMPH ER Tab 5, 10, 15 and 20 mg
- Matching Placebo (Placebo Comparator): Matching Placebo Tablets 5, 10, 15 and 20 mg
  Interventions: Drug: AMPH ER Tab Matching Placebo 5, 10, 15 and 20 mg

INTERVENTIONS:
Drug: AMPH ER Tab 5, 10, 15 and 20 mg — Amphetamine
  Other Names: Amphetamine Extended Release Tablets
  Arms: AMPH ER Tab
Drug: AMPH ER Tab Matching Placebo 5, 10, 15 and 20 mg — Placebo
  Other Names: Amphetamine Extended Release Tablets Matching Placebo
  Arms: Matching Placebo

SUMMARY:
To evaluate the efficacy of AMPH ER TAB compared to placebo in adult patients with ADHD aged 18 to 60 years.

DETAILED DESCRIPTION:
This is a randomized, double-blind (DB), placebo-controlled, parallel, study to assess the efficacy and safety of AMPH ER TAB compared to placebo for the treatment of ADHD in adults aged 18 to 60 years.

After Screening and Baseline evaluations are complete, eligible subjects will be randomized in the study to take DB AMPH ER TAB or matching placebo orally once daily in the morning beginning the day after the Baseline visit for 5 weeks. Dose will be titrated on a weekly basis to reach 20 mg per day. Subjects who cannot tolerate the study drug will be discontinued from the study.

A Math Test placement test will be done at Screening or at Baseline. At Visit 5, efficacy assessments will include the administration of serial Math Tests at pre-dose and at 0.5, 1, 2, 4, 8, 10, 12, 13, and 14 hours post-dose (Primary Endpoint) Adult Investigator Symptom Rating Scale (AISRS) and Clinical Global Impression Scale Severity (CGI-S) will be conducted at Baseline and Visits 1 to 5. Digit Symbol Substitution Test (DSST) will be administered at Baseline and Visit 5 (Secondary Endpoints).

Safety assessments will include treatment-emergent adverse events, physical examination, vital signs, body weight, Columbia Suicide Severity Rating Scale (C-SSRS), and direct questioning to assess for sleep, appetite, mood and psychotic events.

ELIGIBILITY:
Inclusion Criteria

1. Male or female aged 18 to 60 years, inclusive at the time of Screening.
2. Diagnosed with ADHD using the DSM-5 criteria based on the Adults ADHD Clinical Diagnostic Scale (ACDS).
3. IQ within normal range based upon clinical opinion of the Investigator.
4. Baseline AISRS total score greater than or equal to 26.
5. Baseline score of 4 or higher in CGI-S.
6. Females who participate in this study will be of childbearing or non-childbearing potential:

   * Childbearing potential: Physically capable of becoming pregnant
   * Non-childbearing potential:

     * Permanently sterile (i.e., both ovaries removed, uterus removed, or bilateral tubal ligation for at least 6 weeks or documented successful hysteroscopic sterilization); and/or
     * Post-menopausal (no menstrual period for at least 12 consecutive months without any other medical cause).
7. Females of childbearing potential must be non-lactating and must have a negative serum pregnancy test at Screening.
8. Willing to use acceptable, effective methods of contraception.
9. Be able to attend the clinic regularly and reliably.
10. Be able to understand, read, write, and speak English fluently to complete the study related materials.
11. Be informed of the nature of the study and give written consent prior to any study procedure.

Exclusion Criteria:

1. Current or lifetime history of bipolar disorder or any psychotic disorder as established by Mini International Neuropsychiatric Interview (M.I.N.I.) 7.0.2.
2. Current history of major depression, generalized anxiety disorder, obsessive-compulsive disorder, panic disorder, or post-traumatic stress disorder as established by the M.I.N.I. 7.0.2.
3. Known history of chronic medical illnesses including untreated thyroid disease, peripheral vasculopathy, known structural cardiac disorders, serious cardiac conditions, serious arrhythmias, cardiomyopathy, and known family history of sudden death.
4. History of uncontrolled hypertension or a resting systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg. Subjects with well-controlled hypertension on a stable dose for at least 3 months of anti-hypertensives will be allowed to participate.
5. Have clinically significant findings in vital signs measurements at Screening including:

   * Systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg
   * Heart rate >100 bpm
6. Known history or presence of significant renal or hepatic disease, as indicated by clinical laboratory assessment:

   * Liver function test results ≥2 times the upper normal limit
   * Abnormal blood urea nitrogen, or creatinine levels
7. Clinically significant abnormal electrocardiogram or cardiac findings on physical examination (including the presence of a pathologic murmur).
8. Use of the following medications within 14 days of Baseline Visit:

   * Atomoxetine
   * Monoamine oxidase inhibitors (e.g., selegiline, isocarboxazid, phenelzine, tranylcypromine)
   * Tricyclic antidepressants (e.g., desipramine, protriptyline).
9. Use of the following medications within 3 days of Baseline Visit:

   * Gastrointestinal acidifying agents (e.g., guanethidine, reserpine, glutamic acid hydrochloride [HCl], ascorbic acid)
   * Urinary acidifying agents (e.g., ammonium chloride, sodium acid phosphate, methenamine salts).
10. Use of fluoxetine within 30 days of Baseline Visit.
11. Use of stimulant medications within 1 week of Baseline Visit.
12. Planned use of prohibited drugs or agents from the Screening visit through the end of the study.
13. Participation in a clinical study in which an investigational drug was administered within 30 days prior to Screening.
14. Abnormal clinically significant laboratory test values at Screening that, in the opinion of the Medical Monitor or Sponsor, would preclude study participation.
15. Known history of allergy/hypersensitivity to amphetamine or any of the components of AMPH ER TAB.
16. Known history of lack of clinical response to amphetamine based upon Investigator judgment.
17. Positive test result for HIV, Hepatitis B surface antigen, or Hepatitis C antibody.
18. Any uncontrolled medical condition that, in the opinion of Medical Monitor or Sponsor, would preclude study participation.
19. History or presence of alcohol dependence or substance abuse disorder according to DSM-5 or within the last 12 months.
20. Subject's inability or unwillingness to follow directions from the study research staff.
21. Answer of "yes" to questions 4 or 5 of the C-SSRS within the last 2 years.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2019-10-19 (Actual); Study Completion 2019-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J. Cutler, MD, Principal Investigator — Meridien Research Inc.
Locations (3):
- United States (3):
  - Meridien Research, Bradenton, Florida
  - Meridien Research, Inc., Maitland, Florida
  - Center for Psychiatry and Behavioral Medicine, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cutler AJ, Childress AC, Pardo A, Duhoux S, Gomeni R, Rafla E, King TR, Kando JC. Randomized, Double-Blind, Placebo-Controlled, Fixed-Dose Study to Evaluate the Efficacy and Safety of Amphetamine Extended-Release Tablets in Adults With Attention-Deficit/Hyperactivity Disorder. J Clin Psychiatry. 2022 Jul 20;83(5):22m14438. doi: 10.4088/JCP.22m14438. PMID 35857716

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 166 subjects was screened; 36 subjects failed screening. A total of 130 subjects were randomized, 65 to each treatment arm. Three subjects randomized to AMPH ER TAB did not receive drug, resulting in 127 subjects who started the study.
Period: Overall Study
Arm/Group | AMPH ER Tab | Matching Placebo
Started | 62 | 65
Completed | 45 | 46
Not Completed | 17 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AMPH ER Tab | Matching Placebo | Total
Number analyzed (Participants) | 62 | 65 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.1 (11.14) | 31.8 (10.33) | 32.4 (10.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 36 | 76
  Male | 22 | 29 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 36 | 57
  Not Hispanic or Latino | 41 | 29 | 70
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 9 | 16
  White | 52 | 52 | 104
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 62 | 65 | 127

OUTCOME MEASURES:

1. Primary Outcome: Lean Squares Mean (± Standard Error) of Math Test Score Over All Post-dose Time Points (0.5, 1, 2, 4, 8, 10, 12, 13, and 14 Hours Post-dose) Assessed During the Administration of Serial Math Tests at Visit 5 (Week 5)
Description: The Total Math Score is the sum of the number of math problems attempted plus the number of math problems answered correctly and it provides an objective measure of performance that is time-sensitive, ADHD medication-sensitive, and well documented as a measure to evaluate ADHD medication effectiveness throughout the day. The Total Math Score ranges from 0-800 with higher scores indicating better performance.
Time Frame: Pre-dose to 14 hour post-dose
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | AMPH ER Tab | Matching Placebo
Number analyzed (Participants) | 45 | 46
Score on a scale | 259.5 (69.40) | 260.6 (77.75)

2. Secondary Outcome: Change From Baseline in AISRS Total Score at Each Post-baseline Visit
Description: AISRS scale was developed to better capture symptoms of ADHD in adult patients. The scale has 18 items scored as follows: 0 (none), 1 (mild), 2 (moderate), 3 (severe). The maximum total score for the scale is 54 points.
Time Frame: Baseline, Visit 1 (week 1), Visit 2 (week 2), Visit 3 (week 3), Visit 4 (week 4), Visit 5 (week 5)
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | AMPH ER Tab | Matching Placebo
Number analyzed (Participants) | 62 | 62
Score on a scale
  Visit 1 | -7.2 (7.94) | -5.3 (5.95)
  Visit 2 | -11.2 (9.45) | -8.1 (7.22)
  Visit 3 | -15 (9.08) | -8.8 (8.38)
  Visit 4 | -15.4 (10.36) | -9.3 (9.47)
  Visit 5 | -15.9 (10.98) | -9.5 (10.05)

3. Secondary Outcome: Change From Baseline to Visit 5 on DSST
Description: The Digit Symbol Substitution Test (DSST) is a paper-and-pencil cognitive test presented on a single sheet of paper that requires a subject to match symbols to numbers according to a key located on the top of the page. The DSST is sensitive to the presence of cognitive dysfunction as well as to change in cognitive function. The DSST is a 90 second test requiring participants to match symbols with numbers according to a code. Potential scores range from 0 to 100, and lower scores indicate worse performance.
Time Frame: From baseline to week 5
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | AMPH ER Tab | Matching Placebo
Number analyzed (Participants) | 62 | 62
Score on a scale | 4.8 (7.64) | 6.5 (7.21)

4. Secondary Outcome: Change From Baseline on Total Math Test Score Over Each Post-dose Time Points (0.5, 1, 2, 4, 8, 10, 12, 13, and 14 Hours Post-dose) Assessed During the Administration of Serial Math Tests at Visit 5 (Week 5)
Description: as for outcome 1
Time Frame: Visit 5 (week 5)
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | AMPH ER Tab | Matching Placebo
Number analyzed (Participants) | 45 | 46
Score on a scale
  0.5 hours | 64.5 (106.21) | 39.7 (82.74)
  1 hours | 67.9 (107.43) | 27.8 (84.10)
  2 hours | 84.4 (115.37) | 47.0 (84.12)
  4 hours | 81.7 (121.72) | 53.0 (87.84)
  8 hours | 78.8 (121.72) | 48.2 (90.28)
  10 hours | 81.2 (118.64) | 53.8 (85.10)
  12 hours | 85.2 (111.18) | 58.3 (94.97)
  13 hours | 88.8 (120.45) | 47.7 (84.07)
  14 hours | 89 (122.89) | 62.9 (78.34)

5. Secondary Outcome: Change From Baseline in CGI-S Total Score at Each Post-baseline Visit
Description: The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Possible ratings are: 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients.
Time Frame: Baseline, Visit 1 (week 1), Visit 2 (week 2), Visit 3 (week 3), Visit 4 (week 4), Visit 5 (week 5)
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | AMPH ER Tab | Matching Placebo
Number analyzed (Participants) | 62 | 65
Score on a scale
  Visit 1 | -0.6 (0.89) | -0.3 (0.52)
  Visit 2 | -1.0 (1.02) | -0.6 (0.68)
  Visit 3 | -1.3 (1.20) | -0.6 (0.79)
  Visit 4 | -1.4 (1.17) | -0.8 (1.10)
  Visit 5 | -1.3 (1.24) | -0.7 (0.97)

ADVERSE EVENTS:
Time Frame: 5 weeks
Arm/Group | AMPH ER Tab | Matching Placebo
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/65
Other Adverse Events (participants affected / at risk) | 54/62 | 35/65
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AMPH ER Tab (N=62) | Matching Placebo (N=65)
Insomnia (Psychiatric disorders) | 14 | 8
Irritability (Psychiatric disorders) | 11 | 5
Initial insomnia (Psychiatric disorders) | 5 | 3
Anxiety (Psychiatric disorders) | 5 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 30 | 14
Dry Moutn (Gastrointestinal disorders) | 12 | 1
Nausea (Gastrointestinal disorders) | 5 | 2
Headache (Nervous system disorders) | 8 | 4
Dizzines (Nervous system disorders) | 5 | 1
Fatigue (General disorders) | 1 | 4
Tachycardia (Cardiac disorders) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-19): https://cdn.clinicaltrials.gov/large-docs/66/NCT03834766/Prot_SAP_000.pdf